CLINICAL TRIAL: NCT04726397
Title: UNIty-Based MR-Linac Guided AdapTive RadiothErapy for High GraDe Glioma: a Phase 2 Trial (UNITED Trial)
Brief Title: UNIty-Based MR-Linac Guided AdapTive RadiothErapy for High GraDe Glioma: a Phase 2 Trial
Acronym: UNITED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jay Detsky, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3412
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Reduced margin adaptive radiotherapy — Reduced (5 mm) clinical target volume margin with weekly contrast-enhanced adaptive radiation on the MR-Linac treatment machine

SUMMARY:
Glioblastoma (GBM) is a high grade glioma (brain tumor) that is treated with surgery or biopsy followed by radiotherapy (RT) given daily over 3 or 6 weeks with or without an oral chemotherapy. Radiation is targeted to the visible residual tumor on magnetic resonance imaging (MRI) images plus a large margin of 15 to 30 mm to account for possible cancer cells outside the visible tumor and for potential growth or shifts in tumor position throughout the prolonged RT course. Standard RT uses MRI to create a reference plan (with large margins) and treats that same volume every day. This exposes a large amount of healthy brain tissue to radiation leading to toxicity and reduced quality of life.

A new technology, the MR-Linac, combines an MRI scanner and a Linac (radiation delivery machine) into one unit. This allows for "adaptive" RT by obtaining an updated MRI scan each day just prior to treatment, adapting the RT plan to take into account any changes in the tumor or the patient's anatomy on that given day. This allows for a smaller (5 mm) margin on the visible tumor as its position can be tracked daily. The goal of this study is to use adaptive RT with small margins to demonstrate that the local control of the visible tumor is not compromised compared to the large volumes used with standard non-adaptive RT, while determining whether smaller margins lead to decreased radiation toxicity and therefore improved quality of life by minimizing radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Histopathologically confirmed malignant glioma of the brain, Grade 4 (GBM)
* Eligible for RT in 15 or 30 fractions with or without chemotherapy (temozolamide)
* Expected survival greater than 12 weeks
* WHO performance status less than or equal to 2
* Able to converse and answer questionnaires in English language
* Has a maximum final planning volume less than 150 cm3

Exclusion Criteria:

* Contraindications to MRI examination as per standard MRI screening policy
* Contraindication to Gadolinium-based contrast media
* Unable to lie flat in a supine position for 30 minutes
* Poor baseline kidney function with an eGFR < 60 mL/min
* Unable to tolerate immobilization in a head thermoplastic mask
* Patients >140 kg and/or a circumference >60cm
* Previous cranial irradiation
* Infratentorial tumour extent, multifocal of leptomeningeal disease
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Imaging-detected tumor recurrence at the edge of the radiation volume ("marginal" failure) | Within 1 year from end of radiation
  The presence of tumor on contrast-enhanced MRI between 1-2 cm from the edge of the treated radiation volume (commonly known as a marginal failure) within 1 year from radiation.

SECONDARY OUTCOMES:
Tumor volume changes during RT | 6 weeks
  Change in gross tumor volume (%) from start to end of RT
Acute radiation toxicity based on RTOG/EORTC Common Toxicity Criteria | 6 weeks
  Grades 1-4 toxicity during RT in the following categories: skin, CNS, eye, ear, and hematological
Quality of life changes based on EORTC QLQ-C30 | 1 year
  Changes in quality of life during and after RT based on accepted EORTC cancer quality of life instruments administered each week on RT, 1 month post RT, and every 3 months subsequently
Dexamethasone usage | 10 weeks
  Amount of dexamethasone required during RT
Quality of life based on EORTC QLQ-BN20 | 1 year
  Changes in quality of life during and after RT based on accepted EORTC brain tumor quality of life instruments administered each week on RT, 1 month post RT, and every 3 months subsequently

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No